CLINICAL TRIAL: NCT02501356
Title: Effects of ISOThrive on Bodyweight, Body Composition, Hunger/Satiety and Cardiac Risk Measures in Overweight Adults
Acronym: ISOThrive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Griffin Hospital (Other)
Collaborators: ISOThrive Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2014-09
Record Dates: First submitted 2015-04-22; First posted 2015-07-17 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Obesity
Keywords: prebiotic; dietary supplement
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ISOThrive supplement 1 (Active Comparator): Participants assigned to the ISOThrive supplement arm will be provided with daily servings of a supplement for 3 months. Participants will be instructed to take the supplement with water daily, once/day in the morning during the treatment period.
  Interventions: Dietary Supplement: ISOThrive Supplement
- ISOThrive supplement 2 (Active Comparator): Participants assigned to the ISOThrive supplement arm will be provided with daily servings of a supplement for 3 months. Participants will be instructed to take the supplement with water daily, once/day in the morning during the treatment period.
  Interventions: Dietary Supplement: ISOThrive Supplement
- Placebo supplement (Placebo Comparator): Participants assigned to the placebo supplement arm will be provided with daily servings of a supplement for 3 months. Participants will be instructed to take the supplement with water daily, once/day in the morning during the treatment period.
  Interventions: Dietary Supplement: Placebo Supplement

INTERVENTIONS:
Dietary Supplement: ISOThrive Supplement — Consumption of ISOThrive supplements for 3 months
  Arms: ISOThrive supplement 1; ISOThrive supplement 2
Dietary Supplement: Placebo Supplement — Consumption of Placebo supplement (Magnesium stearate or methylcellulose) for 3 months
  Arms: Placebo supplement

SUMMARY:
To compare the effects of daily intake of the ISOThrive supplement vs. a placebo on the primary outcome measure of body weight and secondary outcome measures (hunger/satiety, health-related measures and self-reported quality of life) in a group of overweight but otherwise healthy adults.

DETAILED DESCRIPTION:
Hypothesis

The investigator's hypothesize that daily intake for a 3-month period of the ISOThrive supplement vs. a placebo will demonstrate beneficial effects on the primary outcome measure of body weight and secondary outcome measures (hunger/satiety, health-related measures and self-reported quality of life) in a group of overweight adults.

Specific Aims

* To determine the effects of the ISOThrive supplement on body weight in overweight adults encouraged to reduce calories and exercise regularly, but on an unrestricted diet and without specific exercise instruction. Specifically, to demonstrate a clinically meaningful reduction in body weight in a group of overweight adults after 3 months of daily consumption of the ISOThrive supplement.
* To determine the effects of the ISOThrive supplement on hunger/satiety, body composition, waist circumference, blood pressure, blood glucose levels, blood lipid levels, inflammatory and satiety serum markers and self-reported quality of life in overweight adults encouraged to reduce calories and exercise regularly, but on an unrestricted diet and without specific exercise instruction. Specifically, to demonstrate an improvement in hunger/satiety and a clinically meaningful improvement in other measures in a group of overweight adults after 3 months of daily consumption of the ISOThrive supplement.
* To demonstrate the safety of the ISOThrive supplement in terms of its impact on blood, liver and kidney function in overweight adults. Specifically, to demonstrate the lack of a negative impact on blood, liver and kidney function tests in a group of overweight adults after 3 months of daily consumption of the ISOThrive supplement.
* To determine the effects of the ISOThrive supplement on Gut health. Specifically, to demonstrate improvement in Gut health as measured by abdominal bloating, abdominal gas, and abdominal pain/discomfort at the end of 3 months of daily consumption of the ISOThrive supplement.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 and over and weight not > 350lb
* Age between 18 and 75
* Non-smokers
* Able to read and write in English

Exclusion Criteria:

* Pregnant and/or lactating women
* Evidence or history of substance or alcohol abuse (include if over 5years)
* History of major depression, bipolar disorder or schizophrenia, any type of obsessive-compulsive disorder
* Current history of migraine headaches (include if controlled with medication)
* Current use of any prescription or non-prescription weight loss products
* Tobacco use
* Active eating disorder including anorexia nervosa and bulimia
* Known sensitivity or allergy to any of the ingredients in the product
* Symptomatic coronary artery disease or congestive heart failure
* History of a stroke in the past year
* Symptomatic arrhythmia
* Uncontrolled hypertension (i.e. systolic pressure >180 mmHg and or diastolic > 110 mmHg)
* History of a seizure in the past 5 years
* Any cancer in the past 5 years other than non-melanoma skin cancer or in-situ cervical cancer
* Active or history of inflammatory bowel disease
* Current use of TNF-alpha inhibitor medications
* Current use of COX-2 inhibitor medications
* Current use of JAK inhibitor medications
* History of weight loss procedures including bariatric surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Body Weight | Up to 12 weeks
  Body weight will be measured at the beginning and at the end of the study using a calibrated digital scale.

SECONDARY OUTCOMES:
Hunger/satiety | Up to 12 weeks
  will be assessed at the beginning and at the end of the study using a Visual Analog Scale (VAS) that will ask participants a series of questions to be completed at 2 time points: mid-morning between breakfast and lunch, and late evening between dinner and bed time. The VAS questions require participants to rate on a scale the strength of specific sensations they are feeling (i.e., hunger, thirst, amount of food they could eat "right now", nausea, and fullness) by placing a vertical mark on the scale in response to each question.
Satiety indicators | Up to 12 weeks
  will be assessed at the beginning and end of the study with biological markers using Glucagon-like peptide-1 (GLP-1), PYY and ghrelin.
Dietary intake data | Up to 12 weeks
  Dietary intake will be assessed at the beginning and at the end of the study. Each participant will complete three 24-hour dietary recalls (two for weekdays, and one for a weekend day) using an online Automated Self-Administered 24-Hour Recall (ASA24) (available from the National Cancer Institute at http://riskfactor.cancer.gov/tools/instruments/asa24/). This data will be used to provide a representational measure of intake of kilocalories and macronutrients (protein, fat, and carbohydrates).
Body mass index (BMI) | Up to 12 weeks
  will be measured at the beginning and at the end of the study . BMI will be calculated as weight (kg) divided by height in meters (m) squared. Height will be measured by using a calibrated stadiometer.
Body composition | Up to 12 weeks
  will be measured using bioelectrical impedance analysis, which uses the resistance of electrical flow through the body to estimate body fat. The Tanita SC-240 Body Composition Analyzer will be used to measure body composition. The SC-240 Body Composition Analyzer measures weight and calculates body fat percentage and total body water percentage in addition to BMI. Measures will be taken at baseline, 6 weeks and at the end of the 3-month intervention period.
Leptin | Up to 12 weeks
  Leptin levels will be used as a biomarker to monitor the amount of body fat. Leptin level will be assessed at the beginning and at the end of the study . Leptin is a hormone secreted exclusively by adipose cells in response to an increase in body fat mass, and is an important component in the regulation of long-term hunger and food intake. Leptin serves as the brain's indicator of the body's total energy stores. When leptin levels rise in the bloodstream they bind to receptors in arcuate nucleus (ARC). Leptin suppress the release of neuropeptide Y (NPY), which in turn prevents the release of appetite enhancing hypocretin (orexins) from the lateral hypothalamus. This decreases appetite and food intake, promoting weight loss. It also stimulates the expression of cocaine- and amphetamine-regulated transcript (CART).
Waist circumference | Up to 12 weeks
  will be measured at the beginning and end of the study using guidelines of the National Obesity Expert Panel Report.
Blood pressure | Up to 12 weeks
  will be measured by using a Dinamap Monitor Pro 100 (GE Healthcare, Piscataway, NJ) after sitting for 5 minutes. Both systolic and diastolic pressures will be calculated as the mean value of 2 readings 5 minutes apart for each participant at every time point of assessment. Blood pressure will be assessed at baseline, 6 weeks, and at the end of 3 months
Homeostasis model assessment of insulin resistance (HOMA-IR) | 12 weeks
  will be measured in a fasting state at baseline and 12 weeks. Homeostasis model assessment of insulin resistance (HOMA-IR) values will be calculated from fasting serum glucose and serum insulin levels to gauge the degree of insulin resistance.
Blood Lipid levels | Up to 12 weeks
  Total cholesterol (Tchol), triglycerides (TRIG), and high-density lipoprotein (HDL) will be obtained by direct measurements. Very-low-density lipoprotein (VLDL) and low-density-lipoprotein (LDL) are obtained by calculation: VLDL = TRIG/5; and LDL = Tchol - (VLDL + HDL). The HDL:Tchol ratio will be used to evaluate the impact of the supplement on lipid panel. The lipid profile will be assessed at baseline and at the end of 3 months.
Abdominal symptoms | 12 weeks
  We will assess abdominal bloating, abdominal gas, and abdominal pain/discomfort at 6 weeks and at the end of 3 months. Abdominal symptoms will be assessed using a side effects survey.
Change in Quality of life | Up to 12 weeks
  will be assessed using the SF-12 (http://www.sf-36.org/tools/sf12.shtml). The SF-12v2 Health Survey uses 12 questions to assess 8 domains of health and well-being (general health, physical function, physical role, bodily pain, mental health, emotional role, vitality, and social function) within the past 4 weeks. The SF-12v2 is a practical, reliable, and valid measure of physical and mental health and takes only 2 to 3 minutes to complete. This tool will be administered at baseline and at the end of 3 months.
Liver function | Up to 12 weeks
  will be assessed at baseline and at the end of 3 months via a comprehensive metabolic panel to explore the safety of the ISOThrive supplement. Liver function will be evaluated based on levels of alkaline phosphatase, alanine amino transferase, aspartate amino transferase, and bilirubin.
Kidney function | Up to 12 weeks
  Kidney function will be evaluated using blood urea nitrogen and creatinine.
Urine | Up to 12 weeks
  Urine samples will be collected from participants at baseline and at the end of 3 months. Urinalysis will be used to detect substances or cellular material in the urine associated with different metabolic and kidney disorders.
Complete blood count | Up to 12 weeks
  will be performed to assess the different components of blood.
Stool | Up to 12 weeks
  The stool analysis will be done with samples taken for a subset of 40 subjects. DNA extraction (i.e. purification of DNA from sample), LH-PCR Fingerprinting (i.e to amplify a single copy or a few copies of a piece of DNA across several orders of magnitude, generating thousands to millions of copies of a particular DNA sequence), and Multitag Pyrosequencing (i.e. determining the order of nucleotides in DNA based on the "sequencing by synthesis" principle) will be done with the collected stool at one week before the start of the intervention (i.e. one week before taking product), the day before the start of the intervention, and at the end of 3 months.
Inflammatory biomarkers | Up to 12 weeks
  High sensitivity C-reactive protein, TNF, IL6, IL10 and Interferon gamma will be used to monitor inflammation in our study participants. These biomarkers will be assessed at baseline and at the end of 3 months.
Physical activity | Up to 12 weeks
  Physical activity will be assessed at baseline and at the end of 3 months. PA will be assessed by the International Physical Activity Questionnaire (IPAQ).31 The IPAQ is a valid and reliable tool to assess physical activity in adults. It is a more comprehensive tool containing information on weekly activities in household and yard-work activities, occupational activity, transport, leisure time physical activity and sedentary behavior.

CONTACTS AND LOCATIONS:
Overall Officials: David L. Katz, MD, MPH, Principal Investigator — Yale-Griffin Prevention Research Center; Valentine Y. Njike, MD,MPH, Principal Investigator — Yale-Griffin Prevention Research Center
Locations (1):
- Yale-Griffin Prevention Research Center, Derby, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided